CLINICAL TRIAL: NCT01438294
Title: Effects of Exercise Training on Markers of Lung Inflammation and Clinical Crontrol in Asthma Children
Brief Title: Exercise Training in Asthma Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, PhD, PhD in science Rehabilitation, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASMAPED
Record Dates: First submitted 2011-09-18; First posted 2011-09-22 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Asthma
Keywords: Asthma; childhood; exercise
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Active Comparator): The aerobic training will be done on the treadmill with heart monitors with intensity required to achieve 70% of maximum heart rate reached the maximum test for thirty minutes.
  Interventions: Other: Aerobic exercise group
- Video game (Experimental): The training with video game will be done with heart rate monitors with intensity required to achieve 70% of maximum heart rate reached the maximum test for thirty minutes.Will be used Kinect games ( reflex ridge- Adventure).
  Interventions: Other: Video game group

INTERVENTIONS:
Other: Video game group — The training with video game will be done with heart rate monitors with intensity required to achieve 70% of maximum heart rate reached the maximum test for thirty minutes.Will be used Kinect games ( adventure- reflex ridge).
  Arms: Video game
Other: Aerobic exercise group — A 10 minutes warm up period was performed on a treadmill at 2 km/h prior to each session. After that, exercise training was performed during 30 minutes beginning at 70% of the maximum effort determined in the maximal exercise testing. Before and after each session, 3 measures of the peak flow were performed in the standing position (AssessTM, USA). There was progression in the training intensity throughout the study: if the patient maintained 2 consecutive exercise sessions without symptoms, exercise intensity was increased by 5% of cardiac frequency by using either treadmill speed or grade as previously described (Mendes et al.2011).
  Other Names: treadmill training
  Arms: Aerobic exercise

SUMMARY:
The purpose of this study is to assess the effects of a physical training program with active video game in inflammatory markers, quality of life variables , clinical control and physical and functional respiratory assessment of asthmatic children from 5 to 11 years.

DETAILED DESCRIPTION:
The aim of the present study will be to determine whether an aerobic exercise using an active video game system improves asthma control, lung inflammation and functional capacity in children with moderate or severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5 to 11 years;
* Having a diagnosis of asthma, according to the criteria of the National Heart, Lung, and Blood Institute, and
* Not be included in any program of regular physical activity.

Exclusion Criteria:

* Having received aminophylline and theophylline or oral corticosteroids in the last 30 days;
* Respiratory infection have shown over the past two months;
* Have done with inhaled bronchodilator in less than 12 hours before the assessment;
* Inability to perform any of the tests;
* Have heart disease of inflammatory origin, congenital or ischemic;
* Being in the presence of any infectious process with fever and
* Do not agree to the terms of consent

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelim Leal F DantasGomes, Master, Principal Investigator — University of Nove de Julho; Dirceu Costa, PhD, Study Chair — University of Nove de Julho; Luciana Maria M Sampaio, PhD, Study Director — University of Nove de Julho
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gomes EL, Carvalho CR, Peixoto-Souza FS, Teixeira-Carvalho EF, Mendonca JF, Stirbulov R, Sampaio LM, Costa D. Active Video Game Exercise Training Improves the Clinical Control of Asthma in Children: Randomized Controlled Trial. PLoS One. 2015 Aug 24;10(8):e0135433. doi: 10.1371/journal.pone.0135433. eCollection 2015. PMID 26301706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were randomly allocated to either video game (VGG) or treadmill training (TG) group. 2 sealed envelopes were prepared for each participant, each envelope corresponded to one of the study groups and the envelope was drawn for each participant by the researcher after the baseline measurements have been performed.
Pre-assignment Details: Ten children (7 VGG/3 TG) withdrew from the study: 4 due to changes in the school schedule, 3 abandoned without explanation, 2 due to difficulties in the parents schedule and 1 that moved to another city. Twenty-six patients completed the study (13VGG/13TG).
Groups:
- Video Game: The game "Reflex Ridge" of Kinect Adventure (XBOX 360 KinectTM, Microsoft, USA) was used for training. A 10 minutes warm up period was performed on a treadmill at 2 km/h prior to each session. After that, children played video game, each session lasted 30 minutes and was performed in 10 rounds each one lasting 3 minutes with a 30-second rest interval between rounds. The video game intensity was increased with each round, requiring the child to perform a greater number of jumps, squats, lateral movements and arm movements. Before and after each session, 3 measures of the peak flow were performed in the standing position (AssessTM , USA).
Period: Overall Study
Arm/Group | Aerobic Exercise | Video Game
Started | 16 | 20
Completed | 13 | 13
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Video Game | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (2.0) | 7.5 (1.9) | 7.61 (2.02)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Brazil | 13 | 13 | 26
ACQ6 [Median (Inter-Quartile Range); unit: units on a scale] | 1.16 [0.58 to 1.66] | 1.71 [0.83 to 2.66] | 1.62 [0.58 to 2.66]
FeNO [Mean (Standard Deviation); unit: ppb] | 31.7 (15.73) | 35.5 (19.7) | 33.2 (18.4)
Walked distance [Mean (Standard Deviation); unit: meters] | 607.6 (148.5) | 561.6 (126.9) | 580 (132.4)

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Nitric Oxide (FeNO) Level
Description: The measurement of exhaled FeNO level is performed by several commercially available devices, however the equipment NIOX ® (Aerocrine, Sweden) analyzer is the only FDA-approved and Anvisa (Food and Drug Administration) for clinical monitoring of asthma.
  The measure will be performed before and after the training program of exercise, or pulmonary rehabilitation, by means of portable equipment NIOX MINO ®.
Time Frame: The FeNO level was performed in week 8
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Aerobic Exercise | Video Game
Number analyzed (Participants) | 13 | 13
ppb | 29.3 (21.5) | 23.3 (10.9)

2. Secondary Outcome: Treadmil Test (Bruce Protocol)
Description: A maximal exercise testing was performed in a treadmill using Bruce protocol that has been used to provide information on exercise capacity, physiopathological characteristics during effort, the efficacy of medications and the potential risk for diseases ( Zijp et al. 2010). The test was interrupted when the child reported maximal fatigue or reached the maximum heart rate around 200bpm (Peyer et al. 2011). During the test, blood pressure and peripheral oxygen saturation were quantified and an electrocardiogram was performed. The Borg scale was used to quantify for the sensation of shortness of breath during effort and at rest (Lamb 1995).
  Change from baseline in the distance walked on treadmill test will be consider as outcome measure.
Time Frame: 8 week distance walked on treadmill test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Aerobic Exercise | Video Game
Number analyzed (Participants) | 13 | 13
meters | 895.8 (143.4) | 703.3 (148.3)

3. Secondary Outcome: Body Composition
Description: All participants were evaluated individually, always during the afternoon to avoid circadian changes. Height, weight and abdominal circumference were determined. Tetrapolar bioimpedance was measured using the Biodynamics™ model 310 (Biodynamics Corporation Seattle WA, USA) by positioning the child in the supine position and electrodes in the extremity of the right upper and lower limbs (Goran et al.1993).
Time Frame: baseline and after 8 weeks

4. Secondary Outcome: Pulmonary Function
Description: was performed before and after the inhalation of 400μg of salbutamol (Easy One™, USA), and technical procedures were performed as recommended by ATS/ERS. Predicted normal values were those proposed by Polgar and Promadhat 1971 and a 12% and 200 mL increase in FEV1 from baseline were characterized as a positive response to the bronchodilator) in a climate-controlled room.
Time Frame: baseline and after 8 weeks

5. Other Pre Specified Outcome: Asthma Control Questionnaire (ACQ6) - Clinical Control of Disease
Description: Asthma control questionnaire (ACQ) is a standardized toll to assess clinical control in asthmatic patients and consists of 7 questions, 5 related to asthma symptoms, one regarding the use of short- acting ß2 agonists as rescue medication, and one regarding FEV1 before bronchodilator in percent of predicted.
  ACQ score is the average these items and ranges from 0 (completely controlled) to 6 (uncontrolled) obtained in a 7 days period. The total points is divided by six to provide the final score ( six questions with range 0 to 6 points, maximal 36 points divided by six maximal 6 and mimimal 0)
  The cutoff point for controlled/uncontrolled asthma is 2 points. Patient was classified according ACQ scores into controlled (<0.75), partially controlled (0.75-1.5) and uncontrolled asthma (>1.5). A minimal clinical important difference is 0.5 on a 7-point scale (Juniper et al.2005, Leite et al. 2008 and Ko et al. 2012).
Time Frame: clinical control week 8
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aerobic Exercise | Video Game
Number analyzed (Participants) | 13 | 13
units on a scale | 0.25 [0.08 to 0.50] | 0.25 [0 to 0.58]

6. Other Pre Specified Outcome: Energy Expenditure
Description: Was measured using a biaxial accelerometer (SenseWearTM Pro activity monitor, USA) (Kuys et al. 2011). The equipment was always used on the upper right limb for the determination of skin temperature, galvanic skin response and movement. Energy expenditure was calculated in metabolic equivalents (METS) and calories per minute. The SenseWear arm bandTM was used during the exercise sessions as a comparative parameter of effort intensity in the VGG and TG. The energy expenditure at rest, medium and maximum effort was the average of all sessions of all children.
Time Frame: baseline and during all training sessions 8 weeks

ADVERSE EVENTS:
Arm/Group | Aerobic Exercise | Video Game
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 0/16 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days